CLINICAL TRIAL: NCT00057434
Title: Adjunct Vitamin A Therapy for Tuberculosis and HIV/AIDS
Brief Title: Vitamin A Therapy for Tuberculosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01AI041956-05 (NIH)
Record Dates: First submitted 2003-04-01; First posted 2003-04-03 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2007-08

CONDITIONS: Pulmonary Tuberculosis; HIV Infections
Keywords: Vitamin A
MeSH Terms: conditions — Tuberculosis, Pulmonary; HIV Infections | interventions — Geritol

INTERVENTIONS:
Drug: multivitamin

SUMMARY:
The study will determine whether a daily vitamin and mineral supplement (a multivitamin including Vitamin A) will improve health when added to standard chemotherapy for tuberculosis. This study will compare the effectiveness of the multivitamin in HIV infected and HIV uninfected patients.

DETAILED DESCRIPTION:
By the year 2000, 13.8 % of individuals with HIV will be co-infected with tuberculosis (TB). Despite effective TB chemotherapy, mortality rates remain extremely high, and no simple, inexpensive intervention is available. Prior to the discovery of antibiotic treatment, cod-liver oil, a potent source of Vitamin A, was the standard treatment for TB. Vitamin A is essential for normal immune function, and Vitamin A supplementation is used in many countries to reduce mortality in children. Vitamin A deficiency in HIV infected people has been associated with increased mortality in the United States, Haiti, Malawi, and Uganda. This study will determine whether daily Vitamin A supplementation, given concurrently with TB chemotherapy, will reduce mortality in adults with HIV and TB.

All study participants will receive standard TB chemotherapy (isoniazid, rifampicin, streptomycin, pyrazinamide) for the first 2 months, followed by isoniazid and ethambutol for the following 6 months. Participants will be randomized to receive either a daily vitamin and mineral supplement or placebo. Participants will be followed for 24 months after study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Sputum-confirmed pulmonary tuberculosis
* Resident of Zomba or Blantyre Districts, Malawi
* Willing to take tuberculosis chemotherapy as recommended by the National Tuberculosis Control Programme

Exclusion Criteria:

* Prior treatment for tuberculosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1140
Dates: Start 1998-09

PRIMARY OUTCOMES:
Mortality

SECONDARY OUTCOMES:
Morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Richard D. Semba, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Zomba Central Hospital, Zomba, Malawi

REFERENCES:
- [Derived] Semba RD, Kumwenda J, Zijlstra E, Ricks MO, van Lettow M, Whalen C, Clark TD, Jorgensen L, Kohler J, Kumwenda N, Taha TE, Harries AD. Micronutrient supplements and mortality of HIV-infected adults with pulmonary TB: a controlled clinical trial. Int J Tuberc Lung Dis. 2007 Aug;11(8):854-9. PMID 17705950